CLINICAL TRIAL: NCT03125785
Title: The Effect of Ophthalmic Solutions on Contact Lenses Used After Surgery for Congenital Cataract Investigated in Vivo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Sara De Lima, Optometrist, MSc, St. Erik Eye Hospital
Other Study IDs: saradelima1
Record Dates: First submitted 2017-04-11; First posted 2017-04-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Congenital Cataract
Keywords: congenital cataract, contact lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks

GROUPS / COHORTS (2):
- contact lens and eye drops: Contact lenses collected from patients that have used eye drops containing dexamethasone and benzalkonium chloride for a set period of time and set dosage after surgery
- contact lens and no eye drops: Contact lenses used for the same period of time collected from a control group that has had no surgery and no eye drops in combination with their contact lenses.

SUMMARY:
Patients with congenital cataract operated at St. Erik Eye Hospital are given the topical steroid dexamethasone (Isopto-Maxidex) according to a set treatment plan. They are provided a contact lens made of the polymer Filcon 4A that is frequently replaced due to the results of previous in vitro studies that have shown accumulation of preservatives in the hydrogel contact lens matrix which could question their use in combination with ophthalmic solutions. We conducted a pilot study that indicate that the results in vivo are different from the results in vitro and we suspect that insignificant amounts of dexamethasone and benzalkonium chloride are taken up by the lenses due to tear drainage.

Contact lenses from 30 patients at St. Erik Hospital that have undergone surgery for congenital cataract and are treated with eye drops containing dexamethasone and benzalkonium chloride will be collected and analyzed. Ultraviolet-Visible spectrophotometer (UV-vis) and Laser desorption ionization-mass spectrometry (LDI-MS) will be used to study uptake and release of dexamethasone and benzalkonium chloride. Scanning electron microscopy (SEM) will be used to study surface morphology. Thirty Contact lenses from a control group without topical treatment will also be analyzed. Data will consist of contact lens material, wearing time, pharmaceutical agents, contact lens solution when applicable, diagnosis and possible co-morbidity.

DETAILED DESCRIPTION:
Contact lenses are frequently used as a part of the treatment in professional hospital eye care with indications such as visual aid in keratokonus and scarred corneas and as bandage lenses shielding the cornea in various corneal diseases. An indication of great importance is the providing the visual correction in infants following surgery for congenital cataract. In Sweden, approximately 40 children are born with congenital cataract every year and more than 100 children develop cataract within the first years of life. The cataract can develop in one eye, unilateral cataract, or in both eyes, bilateral cataract. If the cataract is dense it is of great importance to remove the clouded lens as soon as possible to ensure the influx of light and to enable visual development. If the eye is big enough an intraocular lens (IOL) is inserted but if the eye is to small the child is left without an implanted lens. Visual development however requires not only light influx but a sharp image on the retina and to achieve good visual function contact lenses are fitted following surgery. After cataract surgery anti-inflammatory eye drops containing steroids are prescribed for several weeks and the drops are instilled in the eye with the contact lens in place.The effects of eye drops on the contact lenses and possible secondary effects on the eye are largely unknown. The ophthalmic solutions contain active ingredients as well as preservatives such as benzalkonium chloride. Benzalkonium chloride can increase the ocular permeability but also cause irritation at higher concentrations. The uptake of these substances by the lenses can impair the optical clarity of the lenses, cause discoloration, discomfort and irritate the eye. Some studies have shown accumulation of preservatives in the hydrogel contact lens matrix which could question their use in combination with ophthalmic solutions and have led to recommendations of frequent replacement of the lenses. The effects of ophthalmic solutions on the lens materials are not fully understood and most studies are performed in vitro. In collaboration with the Royal Institute of Technology (KTH) methods for measuring drug and preservative uptake by silicone hydrogel contact lenses and to study the surface morphology changes for contact lenses were developed. An in vitro model study showed that active ingredients from eye drops together with preservatives were taken up by the lenses in significant amounts. The method was further implemented in an in vivo pilot study with contact lenses collected from patients treated with different ophthalmologic preparations with the contact lens in place. No traces of active ingredients or preservatives could be found on the worn and treated lenses. The surface morphology changes were minor regardless of the time the lenses were worn or the frequency of medication, which suggests that insignificant amounts of drugs were taken up and the drugs were probably mostly removed by tear drainage. The results are presented in a manuscript that will be sent for publication.

ELIGIBILITY:
Inclusion Criteria:

* Patients that has undergone surgery for congenital cataract
* Must have used contact lenses for 30 +/- days in conjunction with the surgery
* Must have followed the set treatment dexamethasone treatment plan

Exclusion Criteria:

* Patients that has used other eye drops in combination with the investigated drop

Ages: 3 Weeks to 7 Years | Sex: All
Age Groups: Child
Study Population: Contact lenses from children that has undergone surgery for congenital cataract
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Uptake or no uptake of dexamethasone and/or benzalkonium chloride in used contact lenses. | Contact lenses will be collected and analyzed after 30 +/- 5 days of use.
  Contact lenses from patients at St. Erik Eye Hospital that have undergone surgery for congenital cataract and are treated with eye drops containing dexamethasone and benzalkonium chloride will be collected and analyzed. Ultraviolet-Visible spectrophotometer (UV-vis) and Laser desorption ionization-mass spectrometry (LDI-MS) will be used to study uptake and release of dexamthasone and benzalkonium chloride. Scanning electron microscopy (SEM) will be used to study surface morphology. Contact lenses from a control group that has had no surgery and therefore no topical treatment will also be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kugelberg, professor, Study Director — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No